CLINICAL TRIAL: NCT03236116
Title: Almond Consumption and Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Richard Mattes, Professor, Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 055-047
Record Dates: First submitted 2017-07-13; First posted 2017-08-01 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Glucose Intolerance; Appetite Disorders; Glucose Metabolism Disorders (Including Diabetes Mellitus); Lipid Metabolism Disorder
MeSH Terms: conditions — Glucose Intolerance; Feeding and Eating Disorders; Glucose Metabolism Disorders; Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond Group (Experimental): Participants will consumed almonds every day for 6 months, but will not be allowed to consume any other nuts or nut products.
  Interventions: Other: Almonds
- Control Group (Experimental): Participants will continue with their normal eating routine for 6 months, but will not be allowed to consume any nuts or nut products.
  Interventions: Other: Control (no nuts)

INTERVENTIONS:
Other: Almonds — Participants will consume almonds everyday for 6 months.
  Arms: Almond Group
Other: Control (no nuts) — Participants will not be permited to consume any nuts for 6 months.
  Arms: Control Group

SUMMARY:
This study will examine the effects of almonds consumed by adults with different body fat distributions on indices of carbohydrate and lipid metabolism.

DETAILED DESCRIPTION:
There is considerable evidence supporting a causal role for truncal visceral fat depots in glucose dysregulation. Individuals with large visceral fat depots have impaired suppression of free fatty acid release in response to insulin, elevated triglycerides and low concentrations of high density lipoprotein cholesterol. The high free fatty acid concentration may induce insulin resistance in the muscle and liver. There is more recent evidence that truncal subcutaneous fat depots are also problematic, though this literature is mixed. In contrast, gluteo-femoral fat depots have not been implicated in insulin resistance and dysregulation of carbohydrate metabolism. Failure to account for differences in the contributions of these depots will add noise to measurements of dietary interventions to mitigate glucose dysregulation. Previous studies have reported evidence indicating acute and chronic consumption of almonds improves glycemia. Acute effects are important indicators of health benefit, but longer-term trials, ones permitting identification of the effects of a dietary intervention on HbA1c, are more telling and clinically relevant. To more definitively establish the association between almond consumption and improved carbohydrate metabolism, we propose a six-month trial that contrasts the effects of almond consumption at optimal times of the day versus consumption of low nutrient dense snack foods on indices of carbohydrate metabolism, food intake and appetite in adults characterized by three distinct fat depots.

Participants will consume either almonds, or no nuts every day for 6 months. At baseline, participants will be weighed and undergo a DEXA scan to determine body fat composition and will be assigned a group. Blood will also be collected fasted and at stipulated times in response to a meal tolerance test to measure insulin, glucose, C-peptide, HbA1c, lipid panel, gut peptides, and compliance to the diet. Participants will be given links to complete appetite ratings and record food intake. Participants will report to the lab every two weeks to be weighed, and get a resupply of almonds (if in the almond group). At the two-week mark on months 2 and 4, participants will be weighed, blood will be taken to assess compliance to the diet, and links will be given to complete appetite ratings and record food intake. At month 6, all measurements from baseline will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Meeting one of the following body fat distribution criteria determined by DEXA: 1. High visceral fat 2. High gluteo-femoral fat 3. High truncal subcutaneous fat
* 18-60 years
* no nut allergies

Exclusion Criteria:

* Not meeting one of the body fat distribution criteria
* allergic to nuts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline
  HbA1c.
fasting glucose | Baseline
  fasting glucose,
fasting triglycerides | Baseline
  fasting triglycerides
Change in Body weight | Every two weeks for 6 months.
  Body weight
Body composition | Baseline
  Body composition
GLP-1 | Baseline
  GLP-1
Change in HbA1c | 6 months
  HbA1c.
Change in fasting glucose | 6 months
  fasting glucose
fasting triglycerides | 6 months
  fasting triglycerides
Change in Body composition | 6 months
  Body composition
Change in GLP-1 | 6 months
  GLP-1
fasting insulin | Baseline
  fasting insulin
total cholesterol | Baseline
  total cholesterol
LDL-cholesterol | Baseline
  LDL-cholesterol
HDL-cholesterol | Baseline
  HDL-cholesterol
GIP | Baseline
  GIP
change in fasting insulin | 6 months
  fasting insulin
change in total cholesterol | 6 months
  total cholesterol
change in LDL-cholesterol | 6 months
  LDL-cholesterol
change in HDL-cholesterol | 6 months
  HDL-cholesterol
change in GIP | 6 months
  GIP
C-peptide | baseline
C-peptide | 6 months
Homa-IR | baseline
Homa-IR | 6 months
Homa-Percent Beta | Baseline
Homa-Percent Beta | 6 months

SECONDARY OUTCOMES:
Diet Quality | Three days (two non-consecutive week days and one weekend day) at baseline, month 2, 4, and 6.
  Determine the effect of substituting a wholesome snack food (almonds) for more traditional, less nutrient dense, snack foods on total diet quality. Food intake will be measured by the ASA-24 for three days (two non-consecutive week days and one weekend day) at baseline, month 2, 4, and 6.
Compliance | Baseline, month 2, 4, and 6.
  Demonstrate the utility of a novel, sensitive approach to document compliance with a prescription to ingest almonds on a daily basis for six months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Purdue University, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: No